CLINICAL TRIAL: NCT01753570
Title: A Phase 3 Study of MP-424 in Combination With IFN Beta and RBV, in Subjects With Genotype 1/2 Hepatitis C, Who Are Treatment-Naïve or Have Received Interferon Based Therapy
Brief Title: Efficacy and Safety of MP-424, Interferon Beta (IFN Beta), and Ribavirin(RBV) in Treatment-Naïve or Having Received Interferon Based Therapy With Chronic Hepatitis C (CHC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Collaborators: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G060-F1
Record Dates: First submitted 2012-12-13; First posted 2012-12-20 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Chronic Hepatitis C(CHC)
Keywords: Feron
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; Interferon-beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MP-424+RBV+IFN beta, Genotype1 (Experimental)
  Interventions: Drug: MP-424; Drug: RBV(24 weeks); Drug: IFN beta(24 weeks)
- RBV+IFN beta, Genotype1 (Experimental)
  Interventions: Drug: RBV(48 weeks); Drug: IFN beta(48 weeks)
- MP-424+RBV+IFN beta, Genotype2 (Experimental)
  Interventions: Drug: MP-424; Drug: RBV(24 weeks); Drug: IFN beta(24 weeks)

INTERVENTIONS:
Drug: MP-424 — MP-424: 750mg every 8 hours (q8h) for 12 weeks
  Arms: MP-424+RBV+IFN beta, Genotype1; MP-424+RBV+IFN beta, Genotype2
Drug: RBV(24 weeks) — RBV: 600 - 1000mg/day based on body weight for 24 weeks
  Arms: MP-424+RBV+IFN beta, Genotype1; MP-424+RBV+IFN beta, Genotype2
Drug: IFN beta(24 weeks) — IFN beta: 600 MIU/day,6 days/week for initial 4 weeks following to 3 days/week for 24 weeks
  Arms: MP-424+RBV+IFN beta, Genotype1; MP-424+RBV+IFN beta, Genotype2
Drug: RBV(48 weeks) — RBV: 600 - 1000mg/day based on body weight for 48 weeks
  Arms: RBV+IFN beta, Genotype1
Drug: IFN beta(48 weeks) — IFN beta: 600 MIU/day,6 days/week for initial 4 weeks following to 3 days/week for 48 weeks
  Arms: RBV+IFN beta, Genotype1

SUMMARY:
This study will evaluate the efficacy and safety of MP-424 with IFN beta and RBV in patients with genotype 1/2 hepatitis C, who are treatment-naïve or have received its treatment before.

ELIGIBILITY:
Inclusion Criteria:

* Genotype 1 or 2, chronic hepatitis C, with depression(including the past)
* Treatment-naïve(Genotype 1 only) or patient who have ever had previous IFN based treatment
* Able and willing to follow contraception requirements

Exclusion Criteria:

* Cirrhosis of the liver or hepatic failure
* Hepatitis B surface antigen-positive or HIV antibodies-positive
* History of, or concurrent hepatocellular carcinoma
* History of, or concurrent serious depression, schizophrenia, or suicide attempt in the past
* Pregnant, lactating, or suspected pregnant patients, or male patients whose female partner is pregnant

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuoki Kondo, M.D., Study Director — Tanabe Pharma Corporation
Locations (1):
- Toranomon Hospital, Kawasaki, Takatsu-ku, Japan

REFERENCES:
- [Result] Kumada H, Mochida S, Nakamuta M, Suzuki F, Yagi T, Takasaki R, Okai M, Kamiya N, Okada Y, Hirota S, Orihashi M, Ochi M, Chayama K. Efficacy and safety of telaprevir with natural human interferon-beta and ribavirin in Japanese chronic hepatitis C patients with depression. Hepatol Res. 2018 Feb;48(2):184-192. doi: 10.1111/hepr.12914. Epub 2017 Jul 19. PMID 28497489

RESULTS

PARTICIPANT FLOW:
Groups:
- MP-424+RBV+IFN Beta, Genotype1; MP-424+RBV+IFN Beta, Genotype2: Drug: MP-424 MP-424: 750mg every 8 hours (q8h) for 12 weeks Drug: RBV RBV: 600 - 1000 mg/day based on body weight for 24 weeks Drug: IFN beta IFN beta: 600 MIU/day,6 days/week for initial 4 weeks following to 3days /week for 24 weeks
- RBV+IFN Beta, Genotype1: Drug: RBV RBV: 600 - 1000 mg/day based on body weight for 48 weeks Drug: IFN beta IFN beta: 600 MIU/day,6 days/week for initial 4 weeks following to 3days /week for 48 weeks
Period: Overall Study
Arm/Group | MP-424+RBV+IFN Beta, Genotype1 | RBV+IFN Beta, Genotype1 | MP-424+RBV+IFN Beta, Genotype2
Started | 30 | 30 | 14
Completed | 28 | 25 | 13
Not Completed | 2 | 5 | 1
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MP-424+RBV+IFN Beta, Genotype1 | RBV+IFN Beta, Genotype1 | MP-424+RBV+IFN Beta, Genotype2 | Total
Number analyzed (Participants) | 30 | 30 | 14 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (6.4) | 57.6 (10.5) | 55.4 (7.7) | 58.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 9 | 52
  Male | 8 | 9 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Undetectable HCV (Hepatitis C Virus) RNA (Ribonucleic Acid) at 24 Weeks After Completion of Drug Administration (SVR, Sustained Viral Response)
Time Frame: 72 weeks(RBV+IFN beta), 48 weeks(MP-424+RBV+IFN beta)
Measure: Number (95% Confidence Interval); unit: percentage of subjects achieving SVR
Arm/Group | MP-424+RBV+IFN Beta, Genotype1 | RBV+IFN Beta, Genotype1 | MP-424+RBV+IFN Beta, Genotype2
Number analyzed (Participants) | 30 | 30 | 14
percentage of subjects achieving SVR | 63.3 [43.9 to 80.1] | 20.0 [7.7 to 38.6] | 71.4 [41.9 to 91.6]

2. Secondary Outcome: Undetectable HCV RNA at 4 Weeks After Beginning of Drug Administration (RVR, Rapid Viral Response)
Time Frame: 4 weeks
Measure: Number (95% Confidence Interval); unit: percentage of subjects achieving RVR
Arm/Group | MP-424+RBV+IFN Beta, Genotype1 | RBV+IFN Beta, Genotype1 | MP-424+RBV+IFN Beta, Genotype2
Number analyzed (Participants) | 30 | 30 | 14
percentage of subjects achieving RVR | 70.0 [50.6 to 85.3] | 6.7 [0.8 to 22.1] | 92.9 [66.1 to 99.8]

3. Secondary Outcome: Undetectable HCV RNA at Completion of Drug Administration (ETR, End-of-treatment Response)
Time Frame: 48 weeks(RBV+IFN beta), 24 weeks(MP-424+RBV+IFN beta)
Measure: Number (95% Confidence Interval); unit: percentage of subjects achieving ETR
Arm/Group | MP-424+RBV+IFN Beta, Genotype1 | RBV+IFN Beta, Genotype1 | MP-424+RBV+IFN Beta, Genotype2
Number analyzed (Participants) | 30 | 30 | 14
percentage of subjects achieving ETR | 76.7 [57.7 to 90.1] | 30.0 [14.7 to 49.4] | 85.7 [57.2 to 98.2]

4. Secondary Outcome: Undetectable HCV RNA at 12 Weeks After Completion of Drug Administration
Time Frame: 60 weeks(RBV+IFN beta), 36 weeks(MP-424+RBV+IFN beta)
Measure: Number (95% Confidence Interval); unit: percentage of subjects achieving SVR12
Arm/Group | MP-424+RBV+IFN Beta, Genotype1 | RBV+IFN Beta, Genotype1 | MP-424+RBV+IFN Beta, Genotype2
Number analyzed (Participants) | 30 | 30 | 14
percentage of subjects achieving SVR12 | 66.7 [47.2 to 82.7] | 20.0 [7.7 to 38.6] | 71.4 [41.9 to 91.6]

5. Secondary Outcome: Transition of Serum HCV RNA Levels
Time Frame: Baseline，Day2，Day3，1Week，2Weeks，3Weeks，4Weeks，12Weeks，End of treatment，Follow-up 12weeks，Follow-up 24weeks
Population: Participants were excluded from analysis because of dropouts or missing data.
Measure: Median (Inter-Quartile Range); unit: log IU/mL
Arm/Group | MP-424+RBV+IFN Beta, Genotype1 | RBV+IFN Beta, Genotype1 | MP-424+RBV+IFN Beta, Genotype2
Number analyzed (Participants) | 30 | 30 | 14
log IU/mL
  Baseline | 6.73 [6.40 to 7.15] | 6.83 [6.55 to 7.15] | 6.05 [5.45 to 6.75]
  Day2 | 4.15 [3.80 to 4.80] | 5.65 [5.20 to 6.10] | 3.80 [3.10 to 4.40]
  Day3 | 3.35 [3.00 to 3.60] | 4.85 [4.40 to 5.30] | 2.80 [2.30 to 3.30]
  1Week: number analyzed (Participants) | 29 | 29 | 14
  1Week | 2.40 [1.90 to 2.80] | 5.30 [4.50 to 5.70] | 1.25 [0.50 to 2.00]
  2Weeks: number analyzed (Participants) | 29 | 29 | 14
  2Weeks | 1.30 [1.00 to 1.80] | 4.60 [3.70 to 5.30] | 0.50 [0.50 to 1.40]
  3Weeks: number analyzed (Participants) | 28 | 29 | 14
  3Weeks | 0.50 [0.50 to 1.00] | 3.70 [2.90 to 4.80] | 0.50 [0.50 to 0.50]
  4Weeks: number analyzed (Participants) | 28 | 29 | 14
  4Weeks | 0.50 [0.50 to 0.75] | 3.20 [2.00 to 4.20] | 0.50 [0.50 to 0.50]
  12Weeks: number analyzed (Participants) | 24 | 28 | 12
  12Weeks | 0.50 [0.50 to 0.50] | 2.75 [0.50 to 4.75] | 0.50 [0.50 to 0.50]
  End of treatment: number analyzed (Participants) | 29 | 29 | 14
  End of treatment | 0.50 [0.50 to 0.50] | 3.20 [0.50 to 5.60] | 0.50 [0.50 to 0.50]
  Follow-up 12weeks: number analyzed (Participants) | 28 | 25 | 13
  Follow-up 12weeks | 0.50 [0.50 to 6.00] | 6.20 [5.00 to 6.70] | 0.50 [0.50 to 0.50]
  Follow-up 24weeks: number analyzed (Participants) | 28 | 25 | 13
  Follow-up 24weeks | 0.50 [0.50 to 6.60] | 6.20 [5.40 to 6.80] | 0.50 [0.50 to 0.50]

6. Secondary Outcome: Number of Participants With the Emergence of Resistance-associated Variants After MP-424 Administration at the Non-structural 3 Protease Region of HCV.
Description: To examine the emergence of resistance-associated variants after MP-424 administration.
Time Frame: From baseline to 24 weeks after completion of drug administration
Population: "Overall number of participants analyzed" indicates the number of participants who did not achieve SVR and detected HCV RNA as positive at the last visit in each group, MP-424+RBV+IFN Beta, Genotype1 and MP-424+RBV+IFN Beta, Genotype2.
Measure: Number; unit: participants
Arm/Group | MP-424+RBV+IFN Beta, Genotype1 | MP-424+RBV+IFN Beta, Genotype2
Number analyzed (Participants) | 8 | 2
participants
  V36M | 1 | 0
  T54A | 1 | 0
  T54S，A156T，V36A | 1 | 0
  T54A，R155W | 0 | 1
  Not detected | 5 | 1

ADVERSE EVENTS:
Groups:
- MP-424+RBV+IFN Beta, Genotype1; MP-424+RBV+IFN Beta, Genotype2: "Drug: MP-424 MP-424: 750mg every 8 hours (q8h) for 12 weeks Drug: RBV RBV: 600 - 1000 mg/day based on body weight for 24 weeks Drug: IFN beta IFN beta: 600 MIU/day,6 days/week for initial 4 weeks following to 3days /week for 24 weeks
- RBV+IFN Beta, Genotype1: "Drug: RBV RBV: 600 - 1000 mg/day based on body weight for 48 weeks Drug: IFN beta IFN beta: 600 MIU/day,6 days/week for initial 4 weeks following to 3days /week for 48 weeks
Arm/Group | MP-424+RBV+IFN Beta, Genotype1 | RBV+IFN Beta, Genotype1 | MP-424+RBV+IFN Beta, Genotype2
Serious Adverse Events (participants affected / at risk) | 4/30 | 3/30 | 5/14
Other Adverse Events (participants affected / at risk) | 30/30 | 30/30 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MP-424+RBV+IFN Beta, Genotype1 (N=30) | RBV+IFN Beta, Genotype1 (N=30) | MP-424+RBV+IFN Beta, Genotype2 (N=14)
Pneumonia (Infections and infestations) | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1
Optic nerve disorder (Eye disorders) | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MP-424+RBV+IFN Beta, Genotype1 (N=30) | RBV+IFN Beta, Genotype1 (N=30) | MP-424+RBV+IFN Beta, Genotype2 (N=14)
Nasopharyngitis (Infections and infestations) | 8 | 12 | 4
Cystitis (Infections and infestations) | 3 | 1 | 3
Oral herpes (Infections and infestations) | 2 | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 4 | 0
Herpes zoster (Infections and infestations) | 0 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1
Tinea pedis (Infections and infestations) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Acne pustular (Infections and infestations) | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 0 | 1
Eczema impetiginous (Infections and infestations) | 0 | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 25 | 17 | 11
Hyperuricaemia (Metabolism and nutrition disorders) | 7 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 6 | 2 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Insomnia (Psychiatric disorders) | 8 | 6 | 6
Depression (Psychiatric disorders) | 1 | 3 | 1
Abulia (Psychiatric disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 14 | 15 | 6
Dizziness (Nervous system disorders) | 1 | 4 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 2
Tension headache (Nervous system disorders) | 0 | 2 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 1
Pingueculitis (Eye disorders) | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 12 | 6 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 4 | 2
Vomiting (Gastrointestinal disorders) | 4 | 6 | 4
Constipation (Gastrointestinal disorders) | 4 | 6 | 2
Stomatitis (Gastrointestinal disorders) | 4 | 5 | 0
Abdominal discomfort (Gastrointestinal disorders) | 4 | 3 | 4
Gastritis (Gastrointestinal disorders) | 2 | 3 | 0
Cheilitis (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 1 | 1 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 13 | 5 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 8 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 5 | 0 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 4 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 4 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 10 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 3 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Renal disorder (Renal and urinary disorders) | 0 | 0 | 1
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 22 | 26 | 14
Malaise (General disorders) | 18 | 14 | 7
Chills (General disorders) | 1 | 0 | 1
Oedema (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Blood uric acid increased (Investigations) | 13 | 5 | 10
Blood creatinine increased (Investigations) | 12 | 0 | 5
Platelet count decreased (Investigations) | 6 | 11 | 4
Hyaluronic acid increased (Investigations) | 5 | 1 | 2
Blood bilirubin increased (Investigations) | 4 | 2 | 3
Blood triglycerides increased (Investigations) | 4 | 2 | 1
White blood cell count decreased (Investigations) | 3 | 12 | 5
Haemoglobin decreased (Investigations) | 3 | 3 | 1
Neutrophil count decreased (Investigations) | 2 | 9 | 1
Protein urine present (Investigations) | 2 | 4 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 1
Haematocrit decreased (Investigations) | 2 | 0 | 0
Red blood cell count decreased (Investigations) | 2 | 0 | 0
Collagen antigen type IV increased (Investigations) | 2 | 0 | 0
Blood albumin decreased (Investigations) | 1 | 1 | 1
Liver function test abnormal (Investigations) | 1 | 1 | 1
C-reactive protein increased (Investigations) | 1 | 0 | 1
Glucose urine present (Investigations) | 0 | 1 | 1
Blood chloride decreased (Investigations) | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 0 | 1
Thyroid function test abnormal (Investigations) | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1
White blood cells urine positive (Investigations) | 0 | 0 | 1
Neutrophil percentage increased (Investigations) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other